CLINICAL TRIAL: NCT03199638
Title: Exercise Snacks and Glutamine to Improve Glucose Control in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nemours Children's Clinic (Other)
Responsible Party: Principal Investigator, Dominique Darmaun, Principal Investigator, Nemours Children's Clinic
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Nemours IRB #790908
Record Dates: First submitted 2017-06-20; First posted 2017-06-27 (Actual); Results first posted 2023-08-14 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-07

CONDITIONS: Diabetes Mellitus, Type 1; Autoimmune Diseases; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Immune System Diseases; Metabolic Diseases
Keywords: Continuous Glucose Monitoring; Children; Exercise; Glycated hemoglobin; Adolescents; Insulin sensitivity; Glutamine
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Autoimmune Diseases; Diabetes Mellitus; Endocrine System Diseases; Glucose Metabolism Disorders; Immune System Diseases; Metabolic Diseases; Motor Activity; Insulin Resistance | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- an exercise group (Experimental): in which subjects will perform daily 'exercise snacks' within 30 min before breakfast, lunch, and/or dinner or bedtime snack, along with a placebo drink which will be given before breakfast and dinner (twice daily);
  Interventions: Behavioral: Exercise
- an exercise + glutamine group (Experimental): in which subjects will receive a glutamine drink (0.25 g/kg per dose) before breakfast and dinner (twice daily), and perform 'exercise snacks' before each meal
  Interventions: Drug: Glutamine vs. Placebo; Behavioral: Exercise

INTERVENTIONS:
Drug: Glutamine vs. Placebo — oral supplementation with either glutamine or placebo twice daily for 3 months
  Arms: an exercise + glutamine group
Behavioral: Exercise — short bouts of exercise ('exercise snacks') 3 times daily for 3 months

SUMMARY:
This project will assess the feasibility and efficacy of the use of exercise and dietary supplementation with a non essential amino acid - glutamine - a component of most protein supplements, on the regulation of plasma glucose homeostasis in a clinical setting of children with type 1 diabetes (T1D). The study specifically targets patients in puberty as this period is associated with a physiological decline in insulin sensitivity, the latter often associated with poor control. Although physical exercise has long been known to exert beneficial effects on metabolism, lack of time is the most common reason perceived as preventing the performance of exercise in both healthy and diabetic subjects. In earlier studies, the investigators showed that oral supplementation with glutamine, a non essential amino acid given prior to exercise decreases overnight post-exercise blood glucose in adolescents with T1D. Hence, the objective of the current study is to investigate if a novel way of exercising, such as performing 6 short bouts of just 1 min each of intense exercise ('exercise snacks') 30 min before meals, with or without glutamine, improves glycemic control in adolescents with T1D. Designing innovative ways to improve diabetes control in adolescents is highly desirable. The specific aim of the project is to determine whether the sustained use of the proposed exercise snacks with or without glutamine results in diminished glycemic variability and/or improved glucose control

DETAILED DESCRIPTION:
This protocol will help determine whether 'exercise snacks', alone or in combination with dietary glutamine improves diabetes control in adolescents with type 1 diabetes.

All subjects for group A and B will have a full physical exam including Tanner staging as well as waist circumference measurement. A HbA1c, will be obtained as well as fasting triglycerides. A continuous glucose monitor (CGM IPro®, Medtronic Minimed, or a DexCom ^4) will be worn blindly for 6 days and data downloaded. Subjects will then be randomized to 2 study groups of 12 patients each:

(A) an 'exercise group', in which subjects will perform daily 'exercise snacks' within 30 min before breakfast, lunch, and/or dinner or bedtime snack, along with a placebo drink which will be given before breakfast and dinner (twice daily); (B) an 'exercise + glutamine group', in which subjects will receive a glutamine drink (0.25 g/kg per dose) before breakfast and dinner (twice daily), and perform 'exercise snacks' before each meal.

Randomization to the exercise + placebo or the exercise + glutamine group or no exercise+ no glutamine supplements will be stratified according to HbA1c range (eg, 7.0-7.4%; 7.5-8.0 %; 8.4-9.0%;9.5-10%), so as to ensure the comparability of groups.

The placebo and glutamine drink will be prepared at home using measured doses of glutamine or placebo powder to be mixed in a calorie-free, flavored soft drink tailored to the child's individual taste. Patients, families and investigators will be blinded as to the contents of the supplement. Exercise snacks will be designed to be feasible using 6 min worth of simple resistance activities (SRA's) designed by the exercise physiology consultants, Drs. Churilla and Hawley. They may spread them throughout the day if needed. These will consist of activities such as alternating half-squats, calf raises, brief gluteal contractions and knee raises by using stretching bands. The tension of bands may be adjusted as needed during the study. A short video has been created showing the participants how to conduct these exercises and these will be updated periodically in order to keep their interest and compliance. An accelerometer will not be used given the short nature of these bouts of exercise. These will be completed 30 min before breakfast, lunch and dinner.

Patients of group A +B will keep a record of their dietary intake and physical activity for 2 days while CGM is placed (one weekday+ one weekend day) at baseline, during the first week after study initiation and at 1,and 3 months during the study. If the family has a smart phone, a free application will be installed which is "My diet diary calorie count " for better assessment of total caloric intake during this study. Otherwise, a log book would be used. Dietary records will be examined to ensure that potential improvement in glucose control is not due to alterations in dietary intake, such as inadvertently switching to a diet composed of foods with a lower glycemic index. Compliance will be monitored by weekly contact with the study subjects either via phone call or text messaging or via MyNemours. Each participant will also be given a script with the following questions based on the group assignment:

* How many times have you drank your glutamine before meals during the last week?
* How many times have you performed exercise snacks before meals during the last week? In addition, subjects will be asked to check their blood glucose before meals, at bedtime and twice a week around midnight. They will be also asked to record their pulse rate three times weekly at bedtime. A spread sheet will be also provided to each patient for daily documentation of exercise performance and glutamine consumption or text us the results. The number of blood glucose measured per day prior and during the study will be recorded to determine if the compliance with BG checking has increased during the study.

CGM will be placed during the first week after the study initiation, then at one month visit after the enrollment, for 6 days, then all baseline studies, including CGM, HbA1c and triglycerides will be repeated at 3 months. Every patient will undergo a body composition analysis using a dual X-ray absorptiometry (DEXA) at the beginning and the end of the study to express the changes in insulin sensitivity both per kg as well as per kg of fat free mass (FFM).Total insulin dosing will be carefully recorded as units/kg/day during the study.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes for >12 months
* Age between 13 and 19 years
* Males and females at Tanner stage 4 and 5
* All insulin programs, including intermediate,short acting insulin, Lantus, Detemir and short acting insulin or insulin pump therapy.
* Weight of 40 kilograms or higher.
* Hemoglobin A1C between 7%-10% and total daily insulin dose at least 0.9 unit/kg/day.
* BMI between 10 centile to less than 95 percentiles.
* Patients on stable thyroid replacement therapy will be allowed to participate. Exclusion Criteria
* Celiac disease.
* Cystic Fibrosis
* Chronic steroid therapy
* Chronic medications that may interfere with glucose metabolism or liver function.
* History of mental retardation
* Presence of diabetic complications
* Being pregnant or having positive pregnancy test at any time during the study.
* Presence of significant anemia (hemoglobin less than11 g/dL)
* Presence of intercurrent infection
* Subjects involved in an active exercise program or in an organized sport team

Ages: 13 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 14 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Darmaun, PhD, MD, Principal Investigator — Nemours Children's Health System
Locations (1):
- Nemours Children's Clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bloch CA, Clemons P, Sperling MA. Puberty decreases insulin sensitivity. J Pediatr. 1987 Mar;110(3):481-7. doi: 10.1016/s0022-3476(87)80522-x. PMID 2950219
- [Result] Caprio S, Cline G, Boulware S, Permanente C, Shulman GI, Sherwin RS, Tamborlane WV. Effects of puberty and diabetes on metabolism of insulin-sensitive fuels. Am J Physiol. 1994 Jun;266(6 Pt 1):E885-91. doi: 10.1152/ajpendo.1994.266.6.E885. PMID 8023918
- [Result] Amiel SA, Sherwin RS, Simonson DC, Lauritano AA, Tamborlane WV. Impaired insulin action in puberty. A contributing factor to poor glycemic control in adolescents with diabetes. N Engl J Med. 1986 Jul 24;315(4):215-9. doi: 10.1056/NEJM198607243150402. PMID 3523245
- [Result] Arslanian S, Heil BV, Kalhan SC. Hepatic insulin action in adolescents with insulin-dependent diabetes mellitus: relationship with long-term glycemic control. Metabolism. 1993 Mar;42(3):283-90. doi: 10.1016/0026-0495(93)90075-y. PMID 8487645
- [Result] Richter EA, Hargreaves M. Exercise, GLUT4, and skeletal muscle glucose uptake. Physiol Rev. 2013 Jul;93(3):993-1017. doi: 10.1152/physrev.00038.2012. PMID 23899560
- [Result] Wahren J, Felig P, Hagenfeldt L. Physical exercise and fuel homeostasis in diabetes mellitus. Diabetologia. 1978 Apr;14(4):213-22. doi: 10.1007/BF01219419. No abstract available. PMID 640298
- [Result] Goodyear LJ, King PA, Hirshman MF, Thompson CM, Horton ED, Horton ES. Contractile activity increases plasma membrane glucose transporters in absence of insulin. Am J Physiol. 1990 Apr;258(4 Pt 1):E667-72. doi: 10.1152/ajpendo.1990.258.4.E667. PMID 2159218
- [Result] Wasserman DH, Geer RJ, Rice DE, Bracy D, Flakoll PJ, Brown LL, Hill JO, Abumrad NN. Interaction of exercise and insulin action in humans. Am J Physiol. 1991 Jan;260(1 Pt 1):E37-45. doi: 10.1152/ajpendo.1991.260.1.E37. PMID 1987792
- [Result] Baar K, Wende AR, Jones TE, Marison M, Nolte LA, Chen M, Kelly DP, Holloszy JO. Adaptations of skeletal muscle to exercise: rapid increase in the transcriptional coactivator PGC-1. FASEB J. 2002 Dec;16(14):1879-86. doi: 10.1096/fj.02-0367com. PMID 12468452
- [Result] Koopman R, Manders RJ, Zorenc AH, Hul GB, Kuipers H, Keizer HA, van Loon LJ. A single session of resistance exercise enhances insulin sensitivity for at least 24 h in healthy men. Eur J Appl Physiol. 2005 May;94(1-2):180-7. doi: 10.1007/s00421-004-1307-y. Epub 2005 Mar 11. PMID 15761746
- [Result] Silveira AP, Bentes CM, Costa PB, Simao R, Silva FC, Silva RP, Novaes JS. Acute effects of different intensities of resistance training on glycemic fluctuations in patients with type 1 diabetes mellitus. Res Sports Med. 2014;22(1):75-87. doi: 10.1080/15438627.2013.852096. PMID 24392773
- [Result] Davey RJ, Howe W, Paramalingam N, Ferreira LD, Davis EA, Fournier PA, Jones TW. The effect of midday moderate-intensity exercise on postexercise hypoglycemia risk in individuals with type 1 diabetes. J Clin Endocrinol Metab. 2013 Jul;98(7):2908-14. doi: 10.1210/jc.2013-1169. Epub 2013 Jun 18. PMID 23780373
- [Result] Tonoli C, Heyman E, Roelands B, Buyse L, Cheung SS, Berthoin S, Meeusen R. Effects of different types of acute and chronic (training) exercise on glycaemic control in type 1 diabetes mellitus: a meta-analysis. Sports Med. 2012 Dec 1;42(12):1059-80. doi: 10.1007/BF03262312. PMID 23134339
- [Result] Egan AM, Mahmood WA, Fenton R, Redziniak N, Kyaw Tun T, Sreenan S, McDermott JH. Barriers to exercise in obese patients with type 2 diabetes. QJM. 2013 Jul;106(7):635-8. doi: 10.1093/qjmed/hct075. Epub 2013 Mar 23. PMID 23525164
- [Result] Bautista L, Reininger B, Gay JL, Barroso CS, McCormick JB. Perceived barriers to exercise in Hispanic adults by level of activity. J Phys Act Health. 2011 Sep;8(7):916-25. doi: 10.1123/jpah.8.7.916. PMID 21885882
- [Result] Francois ME, Baldi JC, Manning PJ, Lucas SJ, Hawley JA, Williams MJ, Cotter JD. 'Exercise snacks' before meals: a novel strategy to improve glycaemic control in individuals with insulin resistance. Diabetologia. 2014 Jul;57(7):1437-45. doi: 10.1007/s00125-014-3244-6. Epub 2014 May 10. PMID 24817675
- [Result] Mauras N, Xing D, Fox LA, Englert K, Darmaun D. Effects of glutamine on glycemic control during and after exercise in adolescents with type 1 diabetes: a pilot study. Diabetes Care. 2010 Sep;33(9):1951-3. doi: 10.2337/dc10-0275. Epub 2010 Jun 28. PMID 20585005
- [Result] Camera DM, West DW, Phillips SM, Rerecich T, Stellingwerff T, Hawley JA, Coffey VG. Protein ingestion increases myofibrillar protein synthesis after concurrent exercise. Med Sci Sports Exerc. 2015 Jan;47(1):82-91. doi: 10.1249/MSS.0000000000000390. PMID 24870574
- [Result] Stephenson EJ, Lessard SJ, Rivas DA, Watt MJ, Yaspelkis BB 3rd, Koch LG, Britton SL, Hawley JA. Exercise training enhances white adipose tissue metabolism in rats selectively bred for low- or high-endurance running capacity. Am J Physiol Endocrinol Metab. 2013 Aug 1;305(3):E429-38. doi: 10.1152/ajpendo.00544.2012. Epub 2013 Jun 11. PMID 23757406
- [Result] Juvenile Diabetes Research Foundation Continuous Glucose Monitoring Study Group; Tamborlane WV, Beck RW, Bode BW, Buckingham B, Chase HP, Clemons R, Fiallo-Scharer R, Fox LA, Gilliam LK, Hirsch IB, Huang ES, Kollman C, Kowalski AJ, Laffel L, Lawrence JM, Lee J, Mauras N, O'Grady M, Ruedy KJ, Tansey M, Tsalikian E, Weinzimer S, Wilson DM, Wolpert H, Wysocki T, Xing D. Continuous glucose monitoring and intensive treatment of type 1 diabetes. N Engl J Med. 2008 Oct 2;359(14):1464-76. doi: 10.1056/NEJMoa0805017. Epub 2008 Sep 8. PMID 18779236
- [Result] Mauras N, Beck R, Xing D, Ruedy K, Buckingham B, Tansey M, White NH, Weinzimer SA, Tamborlane W, Kollman C; Diabetes Research in Children Network (DirecNet) Study Group. A randomized clinical trial to assess the efficacy and safety of real-time continuous glucose monitoring in the management of type 1 diabetes in young children aged 4 to <10 years. Diabetes Care. 2012 Feb;35(2):204-10. doi: 10.2337/dc11-1746. Epub 2011 Dec 30. PMID 22210571
- [Result] Vilsboll T, Holst JJ. Incretins, insulin secretion and Type 2 diabetes mellitus. Diabetologia. 2004 Mar;47(3):357-366. doi: 10.1007/s00125-004-1342-6. Epub 2004 Feb 13. PMID 14968296
- [Result] Samson SL, Garber A. GLP-1R agonist therapy for diabetes: benefits and potential risks. Curr Opin Endocrinol Diabetes Obes. 2013 Apr;20(2):87-97. doi: 10.1097/MED.0b013e32835edb32. PMID 23403741
- [Result] Weissman PN, Carr MC, Ye J, Cirkel DT, Stewart M, Perry C, Pratley R. HARMONY 4: randomised clinical trial comparing once-weekly albiglutide and insulin glargine in patients with type 2 diabetes inadequately controlled with metformin with or without sulfonylurea. Diabetologia. 2014 Dec;57(12):2475-84. doi: 10.1007/s00125-014-3360-3. Epub 2014 Sep 11. PMID 25208756
- [Result] Ahren B, Johnson SL, Stewart M, Cirkel DT, Yang F, Perry C, Feinglos MN; HARMONY 3 Study Group. HARMONY 3: 104-week randomized, double-blind, placebo- and active-controlled trial assessing the efficacy and safety of albiglutide compared with placebo, sitagliptin, and glimepiride in patients with type 2 diabetes taking metformin. Diabetes Care. 2014 Aug;37(8):2141-8. doi: 10.2337/dc14-0024. Epub 2014 Jun 4. PMID 24898304
- [Result] Rosenstock J, Fonseca VA, Gross JL, Ratner RE, Ahren B, Chow FC, Yang F, Miller D, Johnson SL, Stewart MW, Leiter LA; Harmony 6 Study Group. Advancing basal insulin replacement in type 2 diabetes inadequately controlled with insulin glargine plus oral agents: a comparison of adding albiglutide, a weekly GLP-1 receptor agonist, versus thrice-daily prandial insulin lispro. Diabetes Care. 2014 Aug;37(8):2317-25. doi: 10.2337/dc14-0001. Epub 2014 Jun 4. PMID 24898300
- [Result] Derosa G, Maffioli P. Diabetes: safety and efficacy of albiglutide-results from two trials. Nat Rev Endocrinol. 2014 Sep;10(9):514-6. doi: 10.1038/nrendo.2014.126. Epub 2014 Jul 29. PMID 25069463
- [Result] Prigeon RL, Quddusi S, Paty B, D'Alessio DA. Suppression of glucose production by GLP-1 independent of islet hormones: a novel extrapancreatic effect. Am J Physiol Endocrinol Metab. 2003 Oct;285(4):E701-7. doi: 10.1152/ajpendo.00024.2003. Epub 2003 May 28. PMID 12773303
- [Result] Parlevliet ET, de Leeuw van Weenen JE, Romijn JA, Pijl H. GLP-1 treatment reduces endogenous insulin resistance via activation of central GLP-1 receptors in mice fed a high-fat diet. Am J Physiol Endocrinol Metab. 2010 Aug;299(2):E318-24. doi: 10.1152/ajpendo.00191.2010. Epub 2010 Jun 8. PMID 20530733
- [Result] Greenfield JR, Farooqi IS, Keogh JM, Henning E, Habib AM, Blackwood A, Reimann F, Holst JJ, Gribble FM. Oral glutamine increases circulating glucagon-like peptide 1, glucagon, and insulin concentrations in lean, obese, and type 2 diabetic subjects. Am J Clin Nutr. 2009 Jan;89(1):106-113. doi: 10.3945/ajcn.2008.26362. Epub 2008 Dec 3. PMID 19056578
- [Result] Sherr J, Tsalikian E, Fox L, Buckingham B, Weinzimer S, Tamborlane WV, White NH, Arbelaez AM, Kollman C, Ruedy KJ, Cheng P, Beck RW; Diabetes Research in Children Network. Evolution of abnormal plasma glucagon responses to mixed-meal feedings in youth with type 1 diabetes during the first 2 years after diagnosis. Diabetes Care. 2014 Jun;37(6):1741-4. doi: 10.2337/dc13-2612. Epub 2014 Apr 2. PMID 24696460

RESULTS

PARTICIPANT FLOW:
Groups:
- an Exercise Group,: in which subjects will perform daily 'exercise snacks' within 30 min before breakfast, lunch, and dinner
- Exercise + Glutamine Group: (in which subjects will receive a glutamine drink (0.25g/kg) before breakfast, lunch, and dinner; and perform 'exercise snacks' before each meal.
Period: Overall Study
Arm/Group | an Exercise Group, | Exercise + Glutamine Group
Started | 7 | 7
Completed | 7 | 5
Not Completed | 0 | 2
Not completed — inability to drink glutamine during regularly | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Exercise + Glutamine Group: group performed 'exercise snacks' and received a dietary glutamine supplement
- Exercise Group: group performed 'exercise snacks' only
- Total: Total of all reporting groups
Arm/Group | Exercise + Glutamine Group | Exercise Group | Total
Number analyzed (Participants) | 5 | 7 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 6 | 10
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 17 (1) | 15 (1) | 16 (1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 1 | 4 | 5
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 7 | 12
Height [Mean (Standard Deviation); unit: cm] | 165 (4) | 166 (7) | 165.6 (5.1)
Weight [Mean (Standard Deviation); unit: kg] | 65 (7) | 64 (9) | 64 (8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m²] | 24.0 (2.3) | 23.0 (2.5) | 23.2 (2.4)
BMI percentile [Mean (Standard Deviation); unit: %] | 79 (12) | 78 (12) | 78.5 (11.1)
Duration of diabetes [Mean (Standard Deviation); unit: years] | 6.4 (5.7) | 7.8 (5.1) | 7.2 (5.1)
HbA1C [Mean (Standard Deviation); unit: percentage of total hemoglobin] | 8.3 (0.8) | 7.9 (0.4) | 8.1 (0.6)

OUTCOME MEASURES:

1. Primary Outcome: HbA1c, Glycated Hemoglobin
Description: change in glycated hemoglobin
Time Frame: baseline vs. at 3 months
Measure: Mean (Standard Deviation); unit: percentage of total hemoglobin
Arm/Group | an Exercise Group | an Exercise + Glutamine Group
Number analyzed (Participants) | 7 | 5
percentage of total hemoglobin
  baseline | 7.9 (0.4) | 8.3 (0.8)
  at 3 months | 8.0 (0.6) | 8.4 (0.5)

2. Secondary Outcome: Change in the Mean Amplitude of Glycemic Excursions (MAGE)
Description: MAGE describes the average amplitude of glycemic variations measured using continuous glucose monitoring (CGM)
Time Frame: before vs. at 3 months
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | an Exercise Group | an Exercise + Glutamine Group
Number analyzed (Participants) | 7 | 5
mg/dL
  baseline | 129 (133) | 108 (127)
  at 3 months | 139 (122) | 123 (103)

3. Secondary Outcome: Change in Percent of Blood Glucose (BG) Within Target
Description: Percent of BG between 70 and 180 mg/dL, as measured using Continuous Glucose Monitor (CGM)
Time Frame: baseline vs. at 3 months
Measure: Mean (Standard Deviation); unit: Percentage of Blood Glucose
Arm/Group | an Exercise Group | an Exercise + Glutamine Group
Number analyzed (Participants) | 7 | 5
Percentage of Blood Glucose
  baseline | 63.7 (14.5) | 57.6 (16.8)
  at 3 months | 46.4 (21.1) | 69.2 (18.4)

4. Secondary Outcome: Percent of BG <70 mg/dL
Description: Change in Percent of BG below 70 mg/dL, as determined by Continuous Glucose Monitor (CGM)
Time Frame: baseline vs. at 3 months
Measure: Mean (Standard Deviation); unit: Percentage of Blood Glucose
Arm/Group | an Exercise Group | an Exercise + Glutamine Group
Number analyzed (Participants) | 7 | 5
Percentage of Blood Glucose
  baseline | 7.2 (6.0) | 3.1 (3.1)
  at 3 months | 7.2 (5.1) | 4.4 (2.0)

5. Secondary Outcome: Percent Blood Glucose (BG) >180
Description: Change in Percent of BG above 180 mg, as determined using Continuous Glucose Monitor (CGM)
Time Frame: baseline vs. at 3 months
Measure: Mean (Standard Deviation); unit: Percentage of Blood Glucose
Arm/Group | an Exercise Group | an Exercise + Glutamine Group
Number analyzed (Participants) | 7 | 5
Percentage of Blood Glucose
  basline | 29.1 (15.6) | 39.4 (18.9)
  at 3 months | 46.4 (21.1) | 26.6 (17.8)

6. Secondary Outcome: Insulin Dose
Description: Change in insulin dose (Units/kg/day) used at home
Time Frame: baseline vs. at 3 months
Measure: Mean (Standard Deviation); unit: Units/kg/day
Arm/Group | an Exercise Group | an Exercise + Glutamine Group
Number analyzed (Participants) | 7 | 5
Units/kg/day
  baseline | 1.0 (0.2) | 0.98 (0.1)
  at 3 months | 0.8 (0.1) | 1.0 (0.4)

7. Secondary Outcome: Insulin Sensitivity Score (ISS)
Description: Change in insulin sensitivity score, determined using SEARCH ISS model published equation: logeIS = 4.64725 - 0.02032 × (waist, cm) - 0.09779 × (HbA1c, %) - 0.00235 × (Triglycerides, mg/dL). The range of ISS scores is between 1-15. Higher scores imply a better insulin sensistivity.
Time Frame: baseline vs. at 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | an Exercise Group | an Exercise + Glutamine Group
Number analyzed (Participants) | 7 | 5
score on a scale
  baseline | 2.17 (0.2) | 2.10 (0.19)
  at 3 months | 2.20 (0.17) | 2.16 (0.15)

ADVERSE EVENTS:
Time Frame: 3 months
Groups:
- an Exercise Group,: in which subjects will perform daily 'exercise snacks' within 30 min before breakfast, lunch, and dinner
  No adverse event
- Exercise + Glutamine Group: (in which subjects will receive a glutamine drink (0.25g/kg) before breakfast, lunch, and dinner; and perform 'exercise snacks' before each meal.
  No adverse event
Arm/Group | an Exercise Group, | Exercise + Glutamine Group
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-04-24): https://cdn.clinicaltrials.gov/large-docs/38/NCT03199638/Prot_SAP_000.pdf